CLINICAL TRIAL: NCT04977869
Title: Safety and Efficacy Study of Remote Ischemic Conditioning Combined With Endovascular Thrombectomy for Acute Ischemic Stroke Due to Large Vessel Occlusion of Anterior Circulation: A Multicenter, Randomized, Parallel-controlled Clinical Trial
Brief Title: Safety and Efficacy Study of Remote Ischemic Conditioning Combined With Endovascular Thrombectomy for Acute Ischemic Stroke Due to Large Vessel Occlusion of Anterior Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SERIC-EVT
Record Dates: First submitted 2021-07-13; First posted 2021-07-27 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+Standard medical treatment (Active Comparator): RIC+Standard medical treatment Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 days after endovascular thrombectomy. Additionally, the patients will be treated with standard medical treatment according to the Guidelines for diagnosis and treatment of acute ischemic stroke in China 2018.
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC+Standard medical treatment (Placebo Comparator): Sham RIC+Standard medical treatment Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice daily for 7 days after endovascular thrombectomy. Additionally, the patients will be treated with standard medical treatment according to the Guidelines for diagnosis and treatment of acute ischemic stroke in China 2018.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg.
  Arms: RIC+Standard medical treatment
Procedure: Sham remote ischemic conditioning — Sham remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg.
  Arms: Sham RIC+Standard medical treatment

SUMMARY:
The purpose of this study is to determine the efficacy and safety of remote ischemic conditioning for patients of acute ischemic stroke who underwent endovascular thrombectomy due to large vessel occlusion of anterior circulation.

DETAILED DESCRIPTION:
In this study, 498 cases of ischemic stroke who undergo endovascular thrombectomy within 24 hours from the onset are included in 10 centers in China according to the principle of random, and parallel control. The experimental group receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times per day for 7 consecutive days. The control group receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times per day for 7 consecutive days. Two groups will be followed up for 90 days to evaluate the efficacy and safety of remote ischemic conditioning for patients of acute ischemic stroke who underwent endovascular thrombectomy due to large vessel occlusion of anterior circulation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥ 18 years, male or female
* 2) Diagnosis of acute ischemic stroke within 24 hours of symptom onset and underwent endovascular thrombectomy (EVT) adhering to current guidelines for large vessel occlusion in the anterior circulation (confirmed by computed tomography angiography or digital subtraction angiography)
* 3) Pre-EVT NIHSS ≥ 6
* 4) Premorbid mRS ≤ 2
* 5) Written informed consent obtained from the patient or legally responsible person

Exclusion Criteria:

* 1) Contraindication of endovascular thrombectomy
* 2) Contraindication of remote ischemic conditioning, such as severe soft tissue injury, fracture, or vascular injury in the upper limb, acute or subacute venous thrombosis, arterial occlusive disease, and subclavian steal syndrome
* 3) Head CT showing cerebral hernia and midline displacement
* 4) Pregnancy or lactation
* 5) Previous remote ischemic conditioning therapy or similar treatment
* 6) Severe hepatic and renal dysfunction
* 7) Life expectancy of less than 3 months or inability to complete the study for other reasons
* 8) Unwilling to be followed up or poor compliance
* 9) Current or past participation in other clinical research, or participation in this study within 3 months prior to admission
* 10) Other conditions that the researchers think make the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Scale (mRS) Score 0-2 | 3 months
  Proportion of patients with modified Rankin Scale (mRS) Score 0-2. Ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
National Institute of Health stroke scale (NIHSS) at 24 hours, 7 days (or discharge) after EVT. | 24 hours, 7 days (or discharge)
  National Institute of Health stroke scale (NIHSS) at 24 hours, 7 days (or discharge) after EVT. Ranged from 0 to 42, a low value represents a better outcome.
Barthel Index (BI) at 24 hours, 7 days (or discharge) after EVT. | 24 hours, 7 days (or discharge)
  Barthel Index (BI) at 24 hours, 7 days (or discharge) after EVT. Ranged from 0 to 100, a high value represents a better outcome.
Proportion of patients with modified Rankin Scale (mRS) 0-1 | 90±3 days
  Proportion of patients with modified Rankin Scale (mRS) 0-1. Ranged from 0 to 6, a low value represents a better outcome.
modified Rankin Scale (mRS) score distribution | 90±3 days
  modified Rankin Scale (mRS) score distribution
Recanalization rate within 7 days after EVT | 7 days
  Recanalization rate within 7 days after EVT
Early neurological deterioration at 7 days | 7 days
  Early neurological deterioration at 7 days
Frequency of Hemorrhagic transformation within 7 days | 7 days
  Frequency of Hemorrhagic transformation within 7 days
Frequency of symptomatic intracranial hemorrhage within 7 days | 7 days
  Frequency of symptomatic intracranial hemorrhage within 7 days
Death within 90 days | 90±3 days
  Death within 90 days
Frequency of adverse events within 90 days | 90±3 days
  Frequency of adverse events within 90 days
Adverse events associated with remote ischemic conditioning within 90 days | 90±3 days
  Adverse events associated with remote ischemic conditioning within 90 days
Frequency of serious adverse events within 90 days | 90±3 days
  Frequency of serious adverse events within 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China